CLINICAL TRIAL: NCT06984874
Title: Erector Spinae Plane Block for Children Undergoing Thoracoscopic Sympathectomy: A Prospective Controlled Trial
Brief Title: Erector Spinae Plane Block for Children Undergoing Thoracoscopic Sympathectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, SAFAA MOHAMED SALLAM, Assistant Lecturer of Anesthesiology, Intensive Care and Pain Medicine, Faculty of Medicine, Menoufia University, Egypt., Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/2025
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Erector Spinae Plane Block; Children; Thoracoscopic Sympathectomy
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Experimental): Patients will receive bilateral erector spinae plane block after the induction of general anesthesia as a study group.
  Interventions: Other: Erector spinae plane block
- Control group (Active Comparator): Patients will not receive the block after the induction of general anesthesia as a control group.
  Interventions: Other: General anesthesia

INTERVENTIONS:
Other: Erector spinae plane block — Patients will receive bilateral erector spinae plane block after the induction of general anesthesia as a study group.
  Arms: Erector spinae plane block group
Other: General anesthesia — Patients will not receive the block after the induction of general anesthesia as a control group.
  Arms: Control group

SUMMARY:
This study aims to evaluate the influence of ultrasound-guided erector spinae plane block on postoperative pain and diaphragmatic dysfunction in pediatric patients undergoing thoracoscopic sympathectomy.

DETAILED DESCRIPTION:
Pain may occur after pediatric thoracic surgery in cases such as skin incision creation, rib traction, and drain placement, and in other cases, such as rib nerve injury. Such pain is highly unfavorable to pediatric patients' recovery as it may lead to reduced cough strength for clearing secretions, decreased functional residual capacity, and pulmonary complications such as atelectasis and pneumonia.

Erector spinae plane block (ESPB) is a novel trunk block to relieve chronic neuropathic pain. Since then, it has gained prominence as a regional anesthesia technique with the potential to revolutionize postoperative pain management, and it has been effectively administered not only for the management of perioperative pain for a wide variety of surgeries but also for the management of acute post-traumatic pain and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 to 16 years.
* Either sexes (male or female).
* American Society of Anesthesiologists (ASA) physical status I-II.
* Scheduled for bilateral thoracoscopic sympathectomy under general anesthesia.

Exclusion Criteria:

* History of allergy to local anesthetics.
* Abnormal liver/kidney function.
* Severe spinal deformities.
* Bleeding or coagulation disorders.
* Skin damage or infection at the proposed puncture site.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed on arrival at the post-anesthesia care unit (PACU), 1, 2, 4, 8, 12, and 24 h postoperatively.

SECONDARY OUTCOMES:
Total analgesic consumption | 24 hours postoperatively
  Total analgesic consumption will be recorded.
Anesthetic consumption: minimum alveolar concentration | Intraoperatively
  Anesthetic consumption: minimum alveolar concentration (MAC) of sevoflurane every 10 min using Anesthetic Consumption = Flow Rate × Concentration of Anesthetic in Vapor.
Diaphragmatic excursion | 24 hours postoperatively
  Diaphragmatic excursion will be recorded using ultrasound preoperatively and postoperatively.
Time to the first request for the rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia will be recorded from the end of surgery till first dose of meperidine administrated.
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, and respiratory depression will be recorded.
Recovery profile | 24 hours postoperatively
  Recovery profile will be recorded using Richmond Agitation and Sedation Scale (RASS) was required to be between - 3 and + 4 for a delirium classification (ISMV 4 only; RASS not collected in ISMV 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.